CLINICAL TRIAL: NCT01454596
Title: A Phase I/II Study of the Safety and Feasibility of Administering T Cells Expressing Anti-EGFRvIII Chimeric Antigen Receptor to Patients With Malignant Gliomas Expressing EGFRvIII
Brief Title: CAR T Cell Receptor Immunotherapy Targeting EGFRvIII for Patients With Malignant Gliomas Expressing EGFRvIII
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 110266; 11-C-0266
Record Dates: First submitted 2011-10-06; First posted 2011-10-19 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Malignant Glioma; Glioblastoma; Brain Cancer; Gliosarcoma
Keywords: Cell Therapy; Gene Therapy; Immunotherapy; Brain Cancer; Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — Automobiles; aldesleukin; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I Arm (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + escalating doses of epidermal growth factor receptor (EGFRv)III Chimeric antigen receptor (CAR) transduced peripheral blood lymphocytes (PBL) + aldesleukin
  Interventions: Biological: Epidermal growth factor receptor(EGFRv)III Chimeric antigen receptor (CAR) transduced PBL; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide
- 2/Phase II Arm (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + maximum tolerated dose (MTD) of anti-EGFRvIII CAR transduced PBL established in Phase I + aldesleukin
  Interventions: Biological: Epidermal growth factor receptor(EGFRv)III Chimeric antigen receptor (CAR) transduced PBL; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Epidermal growth factor receptor(EGFRv)III Chimeric antigen receptor (CAR) transduced PBL — Day 0: Cells will be infused intravenously over 20-30 minutes. Patients will receive two cell doses, 2 hours apart.
Drug: Aldesleukin — Aldeskeukin 72,000 IU /kg intravenous (IV) or 720,000 IU /kg IV (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Other Names: Proleukin
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg /m(2)/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg /day X 2 days over 1 hr.
  Other Names: Cytoxan

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with gliomas that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. In this protocol, we are modifying the patient's white blood cells with a retrovirus that has the gene for epidermal growth factor receptor (EGFR) vIII incorporated in the retrovirus.

Objective:

The purpose of this study is to determine a safe number of these cells to infuse and to see if these particular tumor-fighting cells (anti-EGFRvIII cells) are a safe and effective treatment for advanced gliomas.

Eligibility:

- Adults age 18-70 with malignant glioma expressing the EGFRvIII molecule.

Design:

Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed

Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti-EGFRvIII cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}

Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the anti-EGFRvIII cells, and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans every month for the first year, and then every 1-2 months as long as their tumors are shrinking. Follow up visits will take up to 2 days.

DETAILED DESCRIPTION:
BACKGROUND:

- Patients with recurrent gliomas have very limited treatment options. Epidermal growth factor receptor (EGFR).

(EGFRvIII) is the most common mutant variant of EGFR and is present in 24-67% of patients with glioblastoma.

* EGFRvIII expression promotes oncogenesis and is associated with poor prognosis.
* EGFRvIII is not expressed in normal tissue and is an attractive target for immunotherapy.
* We have constructed a retroviral vector that contains a chimeric antigen receptor (CAR) that recognizes the EGFRvIII tumor antigen, which can be used to mediate genetic transfer of this CAR with high efficiency without the need to perform any selection.

OBJECTIVES:

Primary Objectives

* To evaluate the safety of the administration of anti-EGFRvIII CAR engineered peripheral blood lymphocytes in patients receiving the non-myeloablative, lymphodepleting preparative regimen and aldesleukin.
* Determine the six month progression free survival of patients receiving anti-EGFRvIII CAR-engineered peripheral blood lymphocytes and aldesleukin following a nonmyeloablative, lymphodepleting preparative regimen.

ELIGIBILITY:

* Histologically proven glioblastoma or gliosarcoma expressing EGFRvIII as determined by immunohistochemistry (IHC) or Reverse transcription polymerase chain reaction (RT-PCR)
* Failed prior standard treatment with radiotherapy with or without chemotherapy
* Karnofsky performance score (KPS) greater than or equal to 60
* Cardiac, pulmonary and laboratory parameters within acceptable limits

DESIGN:

* The study will be conducted using a Phase I/II design.
* Patients will receive a non-myeloablative, lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumorreactive, CAR gene-transduced peripheral blood mononuclear cells (PBMC), plus intravenous (IV) aldesleukin.
* Once the maximum tolerated cell dose (MTD) has been determined, the study will proceed to the phase II portion.
* In the phase II portion of the trial, patients will be accrued to two cohorts:

  * Patients with recurrent malignant glioma receiving steroids at the time of treatment.
  * Patients with recurrent malignant glioma not receiving steroids at the time of treatment.
* A total of 107 patients may be enrolled over a period of 7 years.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients with histologically proven glioblastomas or gliosarcomas that express epidermal growth factor receptor(EGFRv)III as assessed by immunohistochemistry (IHC) or polymerase chain reaction (PCR) confirmed by the National Cancer Institute (NCI) Laboratory of Pathology.
2. Patients must have progression of disease after radiotherapy (including patients that undergo surgery for recurrent disease and are rendered no evidence of disease (NED)). This includes recurrent glioblastoma (GBM) after receiving all standard first-line treatment, including surgery (if feasible due to neurosurgical and neuro-anatomical considerations) and adjuvant radiotherapy +/- chemotherapy.
3. Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.
4. Age greater than or equal to 18 years and less than or equal to age 70 years.
5. Ability of subject to understand and the willingness to sign a written informed consent document.
6. Willing to sign a durable power of attorney.
7. Karnofsky Performance Status (KPS) greater than or equal to 60
8. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after treatment.
9. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
10. Serology

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by Reverse transcription polymerase chain reaction (RT-PCR) and be Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) negative.
11. Hematology

    * White blood cell (WBC) greater than or equal to 3000/mm(3)
    * Absolute neutrophil count (ANC) greater than or equal to 1000/mm(3) without the support of filgrastim
    * Platelet count greater than or equal to 100,000/mm(3)
    * Hemoglobin greater than or equal to 8.0 g/dl. Subjects may be transfused to reach this cut-off.
12. Chemistry

    * Serum Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) less than or equal to 2.5 x ULN
    * Serum creatinine less than or equal to 1.6 mg/dl
    * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome, who must have a total bilirubin equal to or less than 3.0 mg/dl.
13. Patients must be at least 4 weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide, 3 weeks from procarbazine, 2 weeks from vincristine and 4 weeks from last bevacizumab administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents. All toxicities from prior therapies should be resolved to Common Terminology Criteria in Adverse Events (CTCAE) less than or equal to grade 1 (except for toxicities such as alopecia, or vitiligo).
14. Subject's must be co-enrolled on protocol 03-C-0277

EXCLUSION CRITERIA:

1. A prior history of gliadel implantation in the past six months..
2. Women of child-bearing potential who are pregnant or breast feeding because of the potentially dangerous effects of the treatment on the fetus or infant.
3. Active systemic infections, requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
6. History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
7. History of coronary revascularization or ischemic symptoms.
8. Clinically significant hemorrhagic or ischemic stroke, including transient ischemic attacks and other central nervous system bleeding in the preceding 6 months that were not related to glioma surgery. History of prior intratumoral bleeding is not an exclusion criteria; patients who with history of prior intratumoral bleeding, however, need to undergo a non-contrast head computed tomography (CT) to exclude acute bleeding.
9. Other concomitant anti-cancer therapy except corticosteroids.
10. Any patient known to have left ventricular ejection fraction (LVEF) less than or equal to 45%.
11. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking (greater than or equal to 20 pack-year smoking history, with cessation within the past two years).
    * Symptoms of respiratory dysfunction
12. Patients who are receiving any other investigational agents.
13. Documented LVEF less than or equal to 45% tested in patients:

    * Age greater than or equal to 65 years
    * With clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or have a history of ischemic heart disease and/or chest pain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FRANKEL SA, GERMAN WJ. Glioblastoma multiforme; review of 219 cases with regard to natural history, pathology, diagnostic methods, and treatment. J Neurosurg. 1958 Sep;15(5):489-503. doi: 10.3171/jns.1958.15.5.0489. No abstract available. PMID 13576192
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Bloom HJ. Combined modality therapy for intracranial tumors. Cancer. 1975 Jan;35(1):111-20. doi: 10.1002/1097-0142(197501)35:13.0.co;2-#. PMID 162849
- [Derived] Badhiwala J, Decker WK, Berens ME, Bhardwaj RD. Clinical trials in cellular immunotherapy for brain/CNS tumors. Expert Rev Neurother. 2013 Apr;13(4):405-24. doi: 10.1586/ern.13.23. PMID 23545055
- [Derived] Morgan RA, Johnson LA, Davis JL, Zheng Z, Woolard KD, Reap EA, Feldman SA, Chinnasamy N, Kuan CT, Song H, Zhang W, Fine HA, Rosenberg SA. Recognition of glioma stem cells by genetically modified T cells targeting EGFRvIII and development of adoptive cell therapy for glioma. Hum Gene Ther. 2012 Oct;23(10):1043-53. doi: 10.1089/hum.2012.041. Epub 2012 Sep 24. PMID 22780919
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0266.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients were treated on the Ph I portion of the study. After encountering a patient mortality at dose level 8 and a grade 3 pulmonary toxicity at dose level 9 without seeing any clinical responses, the principal investigator and senior staff re-evaluated the protocol and elected to close the protocol rather than proceed into the Ph II portion.
Groups:
- Group A (Steroids) - Cohort 1: 1x10(7); Group A (Steroids) - Cohort 2: 3x10(7); Group A (Steroids) - Cohort 3: 1x10(8); Group B (No Steroids) - Cohort 1: 1x10(7); Group B (No Steroids) - Cohort 2: 3x10(7); Group B (No Steroids) - Cohort 3: 1x10(8); Group B (No Steroids) - Cohort 4: 3x10(8); Group B (No Steroids) - Cohort 5: 1x10(9): Day 0: Cells will be infused intravenously over 20-30 minutes. Aldeskeukin 72,000 IU /kg intravenous (IV) or 720,000 IU /kg IV (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Days -7 to -3: Fludarabine 25 mg /m(2)/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg /day X 2 days over 1 hr.
- Combined Steroids/no Steroids) - Cohort 6: 3x10(9); Combined Steroids/no Steroids) - Cohort 7: 1x10(10); Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10): After Amendment H, steroid and no steroid groups were no longer separated. Day 0: Cells will be infused intravenously over 20-30 minutes. Aldeskeukin 72,000 IU /kg intravenous (IV) or 720,000 IU /kg IV (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Days -7 to -3: Fludarabine 25 mg /m(2)/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg /day X 2 days over 1 hr.
- Combined Steroids/no Steroids) - Cohort 9: 3x10(10): After Amendment H, steroid and no steroid groups were no longer separated.
  Day 0: Cells will be infused intravenously over 20-30 minutes. Given as a split dose, 2 hours apart.
  Aldeskeukin 72,000 IU /kg intravenous (IV) or 720,000 IU /kg IV (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Days -7 to -3: Fludarabine 25 mg /m(2)/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg /day X 2 days over 1 hr.
Period: Overall Study
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10)
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10) | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 1 | 1 | 17
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 | 43.0 | 52.0 | 46.0 | 57.0 | 56.0 | 53.0 | 55.3 (0.6) | 62.3 (3.2) | 56.0 (11.4) | 47.0 | 57.0 | 54.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Male | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 1 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 3 | 3 | 1 | 1 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1 | 18
Prior Treatment [Count of Participants; unit: Participants] — Procedures/Chemotherapy/Vaccines: Surgery = surg; Radiation = rad; Bevacizumab = beva; Temozolomide = temoz; BCNU = Carmustine; AZD7451 = AZ12607092; EGFRvIII = epidermal growth factor receptor variant III; Vaccine = vacc; Trial = tr; Trebananib = treb; and IMA950 is a vaccine.
  Participants
    Surgery, radiation, temozolomide, bevacizumab,BCNU | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Surgery, radiation, temozolomide, bevacizumab | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
    Surgery, radiation, temozolomide | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 6
    Radiation, temozolomide, bevacizumab | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Surgery,radiation,temozolomide,bevacizumab,AZD7451 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Surgery, radiation, temozolomide, veliparib, beva | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Surg,rad,temozolomide,bevacizumab,EGFRvIII vaccine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Surgery, radiation, temozolomide, IMA950 vaccine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Surg,rad,temoz,EGFRvIIIvacc.vs.placebo tr,bev,treb | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Surgery, radiation, temozolomide, carotuximab,beva | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Surg,rad,temoz,EGFRvIIIvacc.vs.placebo trial,beva | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Related Adverse Events
Description: Aggregate of all adverse events ≥Grade 3 that are possibly, probably, and definitely related to treatment. Adverse events were assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). Per CTCAE, Grade 3 adverse events are severe, Grade 4 is life threatening, and Grade 5 is death.
Time Frame: From 4 weeks after cell infusion up to 77 days
Measure: Number; unit: adverse events
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1
adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

2. Primary Outcome: Progression Free Survival
Description: Progression was assessed by the Response Assessment in Neuro-Oncology (RANO) criteria and is defined as the circumstance when the magnetic resonance imaging (MRI) scan is ranked -2 (definitely worse) or -3 (development of a new lesion).
Time Frame: Time from the date of registration to the date of first observation of progressive disease up to 6 months after end of treatment
Population: Combined steroids/no steroids, Cohort 8: participant experienced a treatment-related mortality (TRM).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1
months | 1.1 | 1.1 | 1.3 | 1.9 | 2.0 | 1.5 | 1.2 | 1.1 [0.9 to 1.3] | 2.7 [0.9 to 12.5] | 1.1 [1.1 to 1.6] | 0 | 2.0

3. Secondary Outcome: Number of Patients With an Objective Response
Description: Objective response was assessed by comparison with baseline dynamic contrast enhanced magnetic resonance imaging with perfusion using Neuro-oncology Working Group proposed guidelines. Complete Response is disappearance of all measurable and non-measurable disease for at least 4 weeks. Partial Response is >/= 50% decrease in lesions for at least 4 weeks. Stable Disease does not meet the criteria for complete response, partial response or progression and requires stable lesions compared with baseline. Progression is >/= 25% increase in lesions.
Time Frame: 4 weeks after cell infusion and monthly as feasible up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Circulating Chimeric Antigen Receptor (CAR+) Cells in Peripheral Blood at 1 Month Post Treatment
Description: CAR and vector presence were quantitated in peripheral blood mononuclear cell (PBMC) samples using established polymerase chain reaction (PCR) techniques
Time Frame: 1 month post transplant
Population: Only 1/3 participants were evaluable in cohort 6 at one month, and 2/3 participants were evaluable in cohort 7 at one month. Due to a low number of events, nonspecific binding of anti-human Fab', and slow recovery of the lymphocyte compartment, the data reported should be interpreted with caution.
Measure: Median (Full Range); unit: K/µL
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 1 | 2 | 1 | 1
K/µL | 23 [23 to 23] | 70 [70 to 70] | 36 [36 to 36] | 67 [67 to 67] | 7 [7 to 7] | 43 [43 to 43] | 28 [28 to 28] | 25 [10 to 219] | 12 [12 to 12] | 67.5 [26 to 109] | NA [NA to NA] — Patient death-data unavailable | 8 [8 to 8]

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 51 dys Grp A, Cohort 1; Cohort 2:68 dys; Cohort 3:40 dys; Grp B, Cohort 1:67 dys; Cohort 2:48 dys; Cohort 3:55 dys; Cohort 4: 46 dys; Cohort 5:147 dys; C. Ster/No Ster Grp, Cohort 6:12 mos, 26 dys; Cohort 7:11 mos, 18 dys; Cohort 8:7 dys; Cohort 9:70 dys.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1
Participants | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 51 days for Group A, Cohort 1; Cohort 2: 68 days; Cohort 3: 40 days; Group B, Cohort 1: 67 days; Cohort 2: 48 days; Cohort 3: 55 days; Cohort 4: 46 days; Cohort 5: 147 days; and Combined Steroids/No Steroids Group, Cohort 6: 12 months and 26 days; Cohort 7: 11 months and 18 days; Cohort 8: 7 days; Cohort 9: 70 days.
Arm/Group | Group A (Steroids) - Cohort 1: 1x10(7) | Group A (Steroids) - Cohort 2: 3x10(7) | Group A (Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 1: 1x10(7) | Group B (No Steroids) - Cohort 2: 3x10(7) | Group B (No Steroids) - Cohort 3: 1x10(8) | Group B (No Steroids) - Cohort 4: 3x10(8) | Group B (No Steroids) - Cohort 5: 1x10(9) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/3 | 0/3 | 0/3 | 1/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/3 | 0/3 | 0/3 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 3/3 | 3/3 | 3/3 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Steroids) - Cohort 1: 1x10(7) (N=1) | Group A (Steroids) - Cohort 2: 3x10(7) (N=1) | Group A (Steroids) - Cohort 3: 1x10(8) (N=1) | Group B (No Steroids) - Cohort 1: 1x10(7) (N=1) | Group B (No Steroids) - Cohort 2: 3x10(7) (N=1) | Group B (No Steroids) - Cohort 3: 1x10(8) (N=1) | Group B (No Steroids) - Cohort 4: 3x10(8) (N=1) | Group B (No Steroids) - Cohort 5: 1x10(9) (N=3) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) (N=3) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) (N=3) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) (N=1) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10) (N=1)
Death not associated with CTCAE term: Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Steroids) - Cohort 1: 1x10(7) (N=1) | Group A (Steroids) - Cohort 2: 3x10(7) (N=1) | Group A (Steroids) - Cohort 3: 1x10(8) (N=1) | Group B (No Steroids) - Cohort 1: 1x10(7) (N=1) | Group B (No Steroids) - Cohort 2: 3x10(7) (N=1) | Group B (No Steroids) - Cohort 3: 1x10(8) (N=1) | Group B (No Steroids) - Cohort 4: 3x10(8) (N=1) | Group B (No Steroids) - Cohort 5: 1x10(9) (N=3) | Combined Steroids/no Steroids) - Cohort 6: 3x10(9) (N=3) | Combined Steroids/no Steroids) - Cohort 7: 1x10(10) (N=3) | Combined Steroids/no Steroids) - Cohort 8: 3-6x10(10) (N=1) | Combined Steroids/no Steroids) - Cohort 9: 3x10(10) (N=1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Pain::Head/headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other (pulmonary edema) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT01454596/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT01454596/ICF_001.pdf